CLINICAL TRIAL: NCT04629599
Title: IPT for Major Depression Following Perinatal Loss: Healing After Loss (HeAL)
Acronym: HeAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Jennifer E. Johnson, C. S. Mott Endowed Professor of Public Health, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD100471 (NIH)
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Perinatal loss; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Interpersonal Psychotherapy; Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal psychotherapy for major depression following perinatal loss (Experimental): Participants in the IPT condition will receive 12 group sessions and 2 individual (pre-group and 1-month booster) sessions as outlined in the manual The individual sessions prepare patients to use the group effectively, to keep group members focused on their treatment goals, and to maintain treatment gains. In addition, 3 of the 12 group sessions will invite women to include their partners or other support people to bolster the woman's social support system and to reduce conflicts over how to react to the loss. These sessions are important because relationship distress is common following perinatal loss. Our IPT intervention allows new women to enter the group every 4 weeks of the 12-week group. Group sessions are semi-structured, and each woman will cover the four group topics three times, approaching each topic from a different stage in the mourning process.
  Interventions: Behavioral: Interpersonal psychotherapy for major depression following perinatal loss
- Coping with Depression (Active Comparator): The Coping with Depression (CWD) course is a structured, manualized psycho-educational group treatment for MDD. The CWD course is based on social learning theory which posits that depression is associated with a decrease in pleasant and an increase in unpleasant person-environment interactions. The problems shown by depressed individuals are viewed as behavioral, with cognitive patterns that can be unlearned or relearned. Its effectiveness is comparable to other forms of psychotherapy in depression. The course content is cognitive-behavioral in nature and is designed to train skills that can be used in the alleviation of depression. The skill modules focus on relaxation, cognitive skills, and behavioral activation. As in the pilot trial, CWD will consist of an individual pregroup session, 12 group therapy sessions (allowing new women to enter every 4th session) and a 1-month individual booster session to provide an identical treatment dose as the experimental condition.
  Interventions: Behavioral: Coping with Depression

INTERVENTIONS:
Behavioral: Interpersonal psychotherapy for major depression following perinatal loss — Participants in the IPT condition will receive 12 group sessions and 2 individual (pre-group and 1-month booster) sessions as outlined in the manual The individual sessions prepare patients to use the group effectively, to keep group members focused on their treatment goals, and to maintain treatment gains. In addition, 3 of the 12 group sessions will invite women to include their partners or other support people to bolster the woman's social support system and to reduce conflicts over how to react to the loss. These sessions are important because relationship distress is common following perinatal loss. Our IPT intervention allows new women to enter the group every 4 weeks of the 12-week group. Group sessions are semi-structured, and each woman will cover the four group topics three times, approaching each topic from a different stage in the mourning process.
  Other Names: IPT
  Arms: Interpersonal psychotherapy for major depression following perinatal loss
Behavioral: Coping with Depression — The Coping with Depression (CWD) course is a structured, manualized psycho-educational group treatment for MDD. The CWD course is based on social learning theory which posits that depression is associated with a decrease in pleasant and an increase in unpleasant person-environment interactions. The problems shown by depressed individuals are viewed as behavioral, with cognitive patterns that can be unlearned or relearned. Its effectiveness is comparable to other forms of psychotherapy in depression. The course content is cognitive-behavioral in nature and is designed to train skills that can be used in the alleviation of depression. The skill modules focus on relaxation, cognitive skills, and behavioral activation. As in the pilot trial, CWD will consist of an individual pregroup session, 12 group therapy sessions (allowing new women to enter every 4th session) and a 1-month individual booster session to provide an identical treatment dose as the experimental condition.
  Other Names: CWD
  Arms: Coping with Depression

SUMMARY:
This study tests the efficacy of interpersonal psychotherapy (IPT) for major depression following perinatal loss (early and late fetal death and early neonatal death) in a sample of 274 women in Flint and Detroit, Michigan. The trial will be the first fully powered randomized trial of treatment for any psychiatric disorder following perinatal loss.

DETAILED DESCRIPTION:
The goal of this study is to conduct a fully-powered randomized efficacy study of IPT for MDD following perinatal loss. Our perinatal-loss adapted group IPT will be compared to a standard depression intervention (CWD, also delivered in a group format) in a sample of 274 women experiencing MDD following perinatal loss. The proposed randomized controlled trial (RCT) will test the hypotheses that: (1) IPT for perinatal loss will result in reduced time to recovery from MDD (primary), depressive symptoms, and PTSD symptoms (secondary) relative to CWD; and that among women meeting criteria for PTSD, IPT will result in reduced time to recovery from PTSD; (2) IPT for perinatal loss will result in increased social support, social role functioning (including parental functioning for women with living children), and well-being, and decreased grief and fear of subsequent pregnancies, relative to CWD; and (3) social support and grief will mediate the effects of IPT on time to MDD recovery.

ELIGIBILITY:
Inclusion Criteria:

* women who meet current Diagnostic and Statistical Manual 5 (DSM-5) criteria for major depressive disorder (MDD)
* have experienced a perinatal loss (including early and late fetal death, death of a liveborn neonate within the first 28 days, and medically recommended termination) within the last 1-12 months
* are 18 to 50 years old
* speak and understand English well enough to understand questionnaires when they are read aloud
* can provide the name and contact information of at least two locator persons
* have access to a telephone through owning one, a relative/friend, or an agency

Exclusion Criteria:

* onset of current major depressive episode prior to news of difficulties with the pregnancy or health risk to the infant (women with prior episodes will be included)
* current or past diagnosis of bipolar disorder, schizophrenia or other psychotic disorder
* primary diagnosis of current substance use disorder
* acute suicidal or homicidal risk
* non-stable course of antidepressant medication or psychotherapy (i.e., beginning or changing dose of either within the previous 12 weeks)
* any IPT or cognitive-behavioral treatment in the previous 12 weeks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult women
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to Major Depressive Disorder recovery | censored at 28 weeks, the proposed study duration
  Assessed via the Longitudinal Interview Follow-up Evaluation (LIFE; lower is better)

SECONDARY OUTCOMES:
Depressive symptoms | 8, 16, and 28 weeks after intake
  Overall score on the Quick Inventory of Depressive Symptoms (QIDS; lower is better)
PTSD symptoms | 8, 16, and 28 weeks after intake
  Life Events Checklist and PTSD Checklist for DSM-5 (LEC-PCL; lower is better)
Time to PTSD recovery | censored at 28 weeks, the proposed study duration
  Assessed via the Longitudinal Interval Follow-Up Evaluation (LIFE; lower is better)
Overall perceived social support | 8, 16, and 28 weeks after intake
  Overall score of the Multidimensional Scale of Perceived Social Support (higher is better)
Dyadic social support (from partner or another important person) | 8, 16, and 28 weeks after intake
  Overall score of the Relationship Assessment Scale (higher is better)
Social role functioning (including parental functioning) | 8, 16, and 28 weeks after intake
  Overall score of the Short version of the Social Adjustment Scale (SAS) - Self Report and parental functioning SAS subscale (lower is better)
Well-being | 8, 16, and 28 weeks after intake
  Overall score of the NIH Neuro-Quality of Life scale for positive affect and well-being (higher is better)
Grief symptoms | 8, 16, and 28 weeks after intake
  Overall score of the Perinatal Bereavement Grief Scale (lower is better)
Complicated grief symptoms | 8, 16, and 28 weeks after intake
  Overall score of the Inventory of Complicated Grief (lower is better)
Perceived deservingness of loss and guilt over loss | 8, 16, an 28 weeks after intake
  Loss Beliefs Scale (lower is better)
Fear of subsequent pregnancies | 8, 16, and 28 weeks after intake
  Overall score of the Fear of subsequent pregnancies measure (lower is better)

OTHER OUTCOMES:
Treatment acceptability | 16 weeks after intake
  Client Satisfaction Questionnaire - Revised (CSQ-8-R; higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Johnson, PhD, Principal Investigator — Michigan State University
Locations (1):
- Anywhere in the entire state of Michigan (treatment is virtual), Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will meet NICHD's timelines and requirements for depositing relevant de-identified data into relevant national databases. This will be reflected in study consent forms. De-identified data will be also made available to qualified researchers upon request, on a compact disk (CD) or other electronic means compatible with our systems. The request will be evaluated by the Principal Investigator to ensure that it meets reasonable standards of scientific integrity.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sharing will occur on NIH-designated timelines.
Access Criteria: Request needs to meet reasonable standards of scientific integrity, as judged by the Study Principal Investigator

REFERENCES:
- [Background] Johnson JE, Price AB, Kao JC, Fernandes K, Stout R, Gobin RL, Zlotnick C. Interpersonal psychotherapy (IPT) for major depression following perinatal loss: a pilot randomized controlled trial. Arch Womens Ment Health. 2016 Oct;19(5):845-59. doi: 10.1007/s00737-016-0625-5. Epub 2016 Mar 22. PMID 27003141
- [Derived] Johnson JE, Price AB, Sikorskii A, Key KD, Taylor B, Lamphere S, Huff C, Cinader M, Zlotnick C. Protocol for the Healing After Loss (HeAL) Study: a randomised controlled trial of interpersonal psychotherapy (IPT) for major depression following perinatal loss. BMJ Open. 2022 Apr 19;12(4):e057747. doi: 10.1136/bmjopen-2021-057747. PMID 35440458